CLINICAL TRIAL: NCT03051035
Title: A Phase 1 First-in-Human Study of KO-947 in Locally Advanced Unresectable or Metastatic, Relapsed and/or Refractory Non-Hematological Malignancies
Brief Title: First-in-Human Study of KO-947 in Non-Hematological Malignancies
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Due to a strategic business decision Kura has stopped development of KO-947. Neither safety nor efficacy reasons were the cause of study termination.
Sponsor: Kura Oncology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KO-ERK-001
Record Dates: First submitted 2017-01-30; First posted 2017-02-13 (Actual); Last update posted 2021-09-20 (Actual); Status verified 2021-09

CONDITIONS: Advanced Malignant Neoplasm
Keywords: non-hematological malignancies; non-squamous; squamous; BRAF; KRAS; NRAS

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- KO-947 (Experimental)
  Interventions: Drug: KO-947

INTERVENTIONS:
Drug: KO-947 — Intravenous administration

SUMMARY:
This phase 1 first-in-human (FIH) dose escalation study will determine the maximum tolerated dose (MTD) of KO-947 in subjects with locally advanced unresectable or metastatic, relapsed and/or refractory, non-hematological malignancies. If an MTD cannot be identified, a recommended phase 2 dose (RP2D) will be determined. In addition, two tumor specific extension cohorts may be conducted to further characterize the safety and tolerability of KO-947 and provide preliminary evidence of anti-tumor activity.

DETAILED DESCRIPTION:
This phase 1 first-in-human (FIH) dose escalation study will determine the maximum tolerated dose (MTD) of KO-947 in subjects with locally advanced unresectable or metastatic, relapsed and/or refractory, non-hematological malignancies. If an MTD cannot be identified, a recommended phase 2 dose (RP2D) will be determined. In addition, two tumor specific extension cohorts may be conducted to further characterize the safety and tolerability of KO-947 and provide preliminary evidence of anti-tumor activity. Three dosing schedules will be executed (Schedule 1, 2, or 3).

Screening evaluations will be completed following signing of informed consent and within either 21 days or 28 days of Cycle 1 Day 1. Evaluations performed as part of the standard of care within 21/28 days of dosing but prior to consent do not need to be repeated. By signing the consent form, study subjects agree to the collection of standard of care health information.

The study will consist of three parts: dose escalation, MTD expansion and tumor specific extension.

ELIGIBILITY:
Key Inclusion Criteria:

1. Subject has a locally advanced unresectable or metastatic, relapsed and/or refractory, non-hematological malignancy for which treatment with an approved agent that is considered standard of care in the indication either does not exist or has proven ineffective.
2. To be enrolled in the dose escalation or in the MTD expansion, Subject must have a locally confirmed diagnosis of either of the following tumor types:

   1. Malignancy of non-squamous histology that carries a BRAF, KRAS, NRAS or HRAS mutation(s).
   2. Malignancy of squamous histology. In cases of mixed histology, squamous must be the predominant histology.
3. Upon the identification of an MTD or RP2D, the Sponsor, in consultation with the study investigators, may open the enrollment of two of the following nonrandomized tumor specific extension cohorts: Subject must have a locally confirmed diagnosis of either of the following tumor types:

   1. RASMUT/BRAFMUT NSCLC: Subject must have a locally confirmed diagnosis of RAS (NRAS, KRAS, HRAS) or BRAF mutated non-small cell malignancies of the lung. Subject must have received at least 1 prior approved regimen for locally advanced or metastatic disease followed by documented progressive disease.
   2. SCCHN and/or SCCE: Subject must have a locally confirmed diagnosis of SCCHN or SCCE with amplification of the 11q13 chromosome. Subject must have received at least 1 prior approved agent for advanced or metastatic disease followed by documented progressive disease. For subjects with 11q13 amplification, the tumor must have >3 copies of the 11q13 chromosome as determined by a methodology approved by the Sponsor.
4. Subject has at least one measurable lesion per RECIST v1.1.
5. For the MTD/RP2D expansion cohort, Subject must have an accessible tumor lesion(s) and consent to tumor biopsy of such a lesion(s) during screening and after starting KO-947 treatment for the analysis of ERK pathway signalling and biological effects.
6. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
7. Serum albumin ≥ 2.8 g/dL
8. Acceptable liver function:

   1. Bilirubin ≤ 1.5 times upper limit of normal (x ULN); if liver metastases are present, then ≤ 2 x ULN is allowed. Criteria does not apply to subjects with Gilbert's syndrome diagnosed as per institutional guidelines.
   2. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 3 x ULN; if liver metastases are present, then ≤ 5 x ULN is allowed.
9. Acceptable renal function with serum creatinine ≤ 1.5 x ULN or a calculated creatinine clearance ≥ 50 mL/min using the Cockcroft-Gault or Modification of Diet in Renal Disease formulas.
10. Acceptable hematologic status:

    1. Absolute neutrophil count (ANC) ≥ 1500 cells/μL
    2. Platelet count ≥ 100,000/μL
    3. Hemoglobin ≥ 9.0 g/dL

Exclusion Criteria:

1. Ongoing treatment with an anticancer agent.
2. History of prior significant toxicity (Grade 2 or higher that required permanent treatment discontinuation) from a BRAF, MEK (MAPK [Mitogen-activated protein]/ERK kinase) or ERK inhibitor.
3. History of retinal vein occlusion, neurosensory retinal detachment, or neovascular macular degeneration. Evidence of visible retinal pathology as assessed by ophthalmologic examination that is considered a risk factor for retinal vein thrombosis or neurosensory retinal detachment.
4. Mean QTcF of >470 ms on triplicate ECGs performed within 5 minutes of each other; subjects currently taking drugs known to be associated with prolonging the QT interval for which there are no adequate therapeutic substitutes; subjects with congenital long QT syndrome. As a guide to known drugs associated with QTc prolongation, please refer to the following Credible Meds web page for a list of drugs that prolong QT and/or cause torsades de pointes, https://crediblemeds.org/pdftemp/pdf/CombinedList.pdf
5. Allergy or hypersensitivity to components of the KO-947 formulation, e.g. dextrose, hydroxypropyl beta cyclodextrin, acetic acid, sodium acetate and water for injection.
6. Participation in any interventional study within 4 weeks of Cycle 1 Day 1 or 5 half-lives of the investigational agent(s) used in the interventional study prior to Cycle 1 Day 1 (whichever is shorter).
7. Grade >1 gastrointestinal toxicity that cannot be managed with supportive care measures.
8. Received treatment for unstable angina within the prior year, myocardial infarction within the prior year, cerebro-vascular attack within the prior year, history of New York Heart Association grade III or greater congestive heart failure, or current serious cardiac arrhythmia requiring medication except atrial fibrillation.
9. Known uncontrolled brain, leptomeningeal or epidural metastases (unless treated and well controlled for at least 4 weeks prior to Cycle 1 Day 1). Controlled brain metastases that require continuous high dose corticosteroid use within 4 weeks of Cycle 1 Day 1.
10. Major surgery, other than diagnostic surgery, within 4 weeks prior to Cycle 1 Day 1, without complete recovery.
11. Active, uncontrolled bacterial, viral, or fungal infections, requiring systemic therapy. Known infection with human immunodeficiency virus, or an active infection with hepatitis B or hepatitis C.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2017-04-06 (Actual); Primary Completion 2020-06-02 (Actual); Study Completion 2020-06-02 (Actual)

PRIMARY OUTCOMES:
To determine the maximal tolerated dose (MTD) and/or the recommended Phase 2 dose (RP2D) of KO-947 in subjects with locally advanced unresectable or metastatic, relapsed and/or refractory, non-hematological malignancies. | Dose-limiting toxicities will be evaluated during the first 28 days of KO-947 monotherapy treatment in the dose escalation portion of the study.

SECONDARY OUTCOMES:
Number of patients that experience Adverse Events (AEs) | Until 30 days after the end of study
  Adverse Events (AEs) and Serious Adverse Events (SAEs) will be graded according to the NCI-CTCAE (Version 4.03)
Maximum plasma concentration (Cmax) of KO-947 on Cycle 1 Day 1 and Cycle 2 Day 1 | Blood samples for determination of KO-947 concentration will be collected at 0, 1, end of infusion, 1.5 2, 2.5 3, 3.5, 4, 6, 8, 24 hours during dose escalation and dose expansion.
Plasma concentration of KO-947 over 24 hours after dosing on Cycle 1 Day 1 and Cycle 2 Day 1 | Blood samples for determination of KO-947 concentration will be collected at 0, 1, end of infusion, 1.5 2, 2.5 3, 3.5, 4, 6, 8, 24 hours during dose escalation and dose expansion.
Time to maximum plasma concentration (tmax) of KO-947 on Cycle 1 Day 1 and Cycle 2 Day 1 | Blood samples for determination of KO-947 concentration will be collected at 0, 1, end of infusion, 1.5 2, 2.5 3, 3.5, 4, 6, 8, 24 hours during dose escalation and dose expansion.
Time to the last detectable plasma concentration (tlast) of KO-947 on Cycle 1 Day 1 and Cycle 2 Day 1 | Blood samples for determination of KO-947 concentration will be collected at 0, 1, end of infusion, 1.5 2, 2.5 3, 3.5, 4, 6, 8, 24 hours during dose escalation and dose expansion.
Terminal half-life (t½λz) of KO-947 on Cycle 1 Day 1 and Cycle 2 Day 1 | Blood samples for determination of KO-947 concentration will be collected at 0, 1, end of infusion, 1.5 2, 2.5 3, 3.5, 4, 6, 8, 24 hours during dose escalation and dose expansion.
Area under the plasma concentration-time curve for KO-947 from zero to 24 hours [AUC(0-24)] on Cycle 1 Day 1 and Cycle 2 Day 1 | Blood samples for determination of KO-947 concentration will be collected at 0, 1, end of infusion, 1.5 2, 2.5 3, 3.5, 4, 6, 8, 24 hours during dose escalation and dose expansion.
Area under the plasma concentration-time curve for KO-947 from zero to the last detectable plasma concentration [AUC(0-last)] on Cycle 1 Day 1 and Cycle 2 Day 1 | Blood samples for determination of KO-947 concentration will be collected at 0, 1, end of infusion, 1.5 2, 2.5 3, 3.5, 4, 6, 8, 24 hours during dose escalation and dose expansion.
Trough plasma concentration (Ctrough) of KO-947 on Cycle 1 Day 1 and Cycle 2 Day 1 | Blood samples for determination of KO-947 concentration will be collected at 0, 1, end of infusion, 1.5 2, 2.5 3, 3.5, 4, 6, 8, 24 hours during dose escalation and dose expansion.
Objective Response Rate (ORR), Progression Free Survival (PFS) and Duration of Response (DOR) of KO-947 | 36 months (approximately 24 months accrual + 12 months follow-up)
  Tumor assessments will be performed approximately every 12 weeks (Schedules 1 and 2) or every 9 weeks (Schedule 3) until disease progression.

CONTACTS AND LOCATIONS:
Locations (5):
- United States (3):
  - Mayo Clinic, Rochester, Minnesota
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
- Spain (2):
  - Vall D'Hebron Institute of Oncology, Barcelona
  - START Madrid-HM CIOCC, Madrid

IPD SHARING:
Plan to Share IPD: Undecided